CLINICAL TRIAL: NCT03606681
Title: Evaluation of Indirect Pulp Capping in Children With Different Materials
Brief Title: Clinical and Radiographic Evaluation of Indirect Pulp Capping in Primary and Permanent Teeth With Different Materials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Altinbas University (Other)
Collaborators: Istanbul University (Other)
Responsible Party: Principal Investigator, Aliye Tugce Gurcan, Assist. Prof., Altinbas University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 35793
Record Dates: First submitted 2018-07-02; First posted 2018-07-31 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Dental Pulp Capping
Keywords: Dental Pulp; calcium hydroxide; Dental Pulp Capping
MeSH Terms: interventions — Calcium Hydroxide; Dycal; Pulp Capping and Pulpectomy Agents; mineral trioxide aggregate; ProRoot MTA

STUDY DESIGN:
Oversight: FDA-regulated Drug: No

ARMS (3):
- Calcium Hydroxide (Dycal) (Active Comparator): Indirect pulp capping treatment with Calcium Hydroxide
  Interventions: Drug: Calcium Hydroxide; Drug: Mineral Trioxide Aggregate; Drug: TheraCal LC
- Mineral Trioxide Aggregate (ProRoot MTA) (Experimental): Indirect pulp capping treatment with Mineral Trioxide Aggregate
  Interventions: Drug: Calcium Hydroxide; Drug: Mineral Trioxide Aggregate; Drug: TheraCal LC
- Theracal LC (Experimental): Indirect pulp capping treatment with Theracal LC
  Interventions: Drug: Calcium Hydroxide; Drug: Mineral Trioxide Aggregate; Drug: TheraCal LC

INTERVENTIONS:
Drug: Calcium Hydroxide — After cleaning the caries with partial removal (non-exposed pulp), cavity disinfected with sodium hypochlorite then indirect pulp capping agent was applied to cavity and restoration was finished in the same session.
  Other Names: Dycal; Pulp capping agent
Drug: Mineral Trioxide Aggregate — After cleaning the caries with partial removal (non-exposed pulp), cavity disinfected with sodium hypochlorite then indirect pulp capping agent was applied to cavity and restoration was finished in in the same session.
  Other Names: (ProRoot MTA)
Drug: TheraCal LC — After cleaning the caries with partial removal (non-exposed pulp), cavity disinfected with sodium hypochlorite then indirect pulp capping agent was applied to cavity (2 milimeter layer) and polymerized and restoration was finished in in the same session.
  Other Names: resin-based calcium silicate cement

SUMMARY:
Indirect pulp capping (IPC) is a treatment that preserves pulp's vitality. Several materials have been used for this procedure. The aim of this study is to evaluate the radiographic and clinical outcomes of TheraCal LC (Bisco Inc., Schaumburg, IL, USA) and to compare it with mineral trioxide aggregate (MTA) (Pro Root MTA, Dentsply Tulsa, Johnson City, TN, USA) and calcium hydroxide [Ca(OH)2] (Dycal, Dentsply De Trey Konstanz, Germany) biomaterials in IPC treatment.

DETAILED DESCRIPTION:
A total of 295 teeth, including second primary molars and first permanent molars with IPC indications from healthy and cooperative children between the ages of 4-15, were included in this study. Teeth were divided into three groups according to the materials used for pulp capping. Indirect pulp treatment was applied using Dycal for 91 teeth, ProRoot MTA for 89 teeth and TheraCal LC for 115 teeth. Primary molars were restored with the compomer material, and permanent molars were restored with the resin composite material. Restorations were evaluated with the Modified United States Public Health Service (modified USPHS) criteria. Clinical and radiographic findings were evaluated for 24 months at follow-up.

ELIGIBILITY:
Inclusion Criteria:

* teeth with clinical and radiographical indications of indirect pulp capping
* systemically healthy and cooperative children

Exclusion Criteria:

* teeth with contraindications of indirect pulp capping: Clinical Exclusion Criteria
* Pain (spontaneous and chronic)
* Fistula
* Acute pulpal inflammation
* Pain with percussion
* Pathologic mobility
* Abscess
* Devitality symptoms (negative response to thermal pulp test) Radiographic Exclusion Criteria
* Progression of caries lesion to pulp
* Perforation of pulp
* Intermittent or irregular lamina dura
* Expanded range of periodontal ligament
* Periapical radiolucency
* Internal and external resorption
* systemically unhealthy and uncooperative children

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Clinical success rates of the indirect pulp capping biomaterials | 24 months
  No pathological symptom like abscess, fistulas or pain at percussion

SECONDARY OUTCOMES:
Success rates according to Modified USPHS criterias | 24 months
  No failed restorations during the controls
Radiographical success rates of the indirect pulp capping biomaterials | 24 months
  No radiolucency or root resorption, healing with dentin bridge

CONTACTS AND LOCATIONS:
Overall Officials: Aliye Tuğçe Gürcan, Assist.Prof., Principal Investigator — Altinbas University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fuks AB. Vital pulp therapy with new materials for primary teeth: new directions and treatment perspectives. J Endod. 2008 Jul;34(7 Suppl):S18-24. doi: 10.1016/j.joen.2008.02.031. PMID 18565366
- [Background] Marchi JJ, de Araujo FB, Froner AM, Straffon LH, Nor JE. Indirect pulp capping in the primary dentition: a 4 year follow-up study. J Clin Pediatr Dent. 2006 Winter;31(2):68-71. doi: 10.17796/jcpd.31.2.y4um5076341226m5. PMID 17315796
- [Background] Gruythuysen RJ, van Strijp AJ, Wu MK. Long-term survival of indirect pulp treatment performed in primary and permanent teeth with clinically diagnosed deep carious lesions. J Endod. 2010 Sep;36(9):1490-3. doi: 10.1016/j.joen.2010.06.006. PMID 20728715
- [Background] Gandolfi MG, Siboni F, Prati C. Chemical-physical properties of TheraCal, a novel light-curable MTA-like material for pulp capping. Int Endod J. 2012 Jun;45(6):571-9. doi: 10.1111/j.1365-2591.2012.02013.x. Epub 2012 Mar 31. PMID 22469093
- [Background] Kotsanos N, Arizos S. Evaluation of a resin modified glass ionomer serving both as indirect pulp therapy and as restorative material for primary molars. Eur Arch Paediatr Dent. 2011 Jun;12(3):170-5. doi: 10.1007/BF03262801. PMID 21640064
- [Background] Al-Zayer MA, Straffon LH, Feigal RJ, Welch KB. Indirect pulp treatment of primary posterior teeth: a retrospective study. Pediatr Dent. 2003 Jan-Feb;25(1):29-36. PMID 12627699
- [Background] George V, Janardhanan SK, Varma B, Kumaran P, Xavier AM. Clinical and radiographic evaluation of indirect pulp treatment with MTA and calcium hydroxide in primary teeth (in-vivo study). J Indian Soc Pedod Prev Dent. 2015 Apr-Jun;33(2):104-10. doi: 10.4103/0970-4388.155118. PMID 25872627
- [Background] Casagrande L, Bento LW, Dalpian DM, Garcia-Godoy F, de Araujo FB. Indirect pulp treatment in primary teeth: 4-year results. Am J Dent. 2010 Feb;23(1):34-8. PMID 20437725